CLINICAL TRIAL: NCT05969665
Title: Effect of Monitoring Continuous Glucose Levels and Physical Activity Via Wearables on Cardiovascular Risk Factors After Cardiac Rehabilitation - A Randomised Controlled Trial: MITIGATE-RF
Brief Title: Effect of Monitoring Continuous Glucose Levels and Physical Activity Via Wearables on Cardiovascular Risk Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-D0040; kt23vanderstouwe
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Coronary Heart Disease; Physical Activity; Cardiovascular Risk Factors
Keywords: blood pressure; lipids; glucose level; smoking; weight; diet
MeSH Terms: conditions — Coronary Disease; Motor Activity; Smoking; Body Weight

STUDY DESIGN:
Intervention Model Description: single-centre, randomized controlled, open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearing a smartwatch and glucose measuring device (Experimental): The intervention will be wearing a smart watch as well as continuous glucose monitoring with direct feedback via an application. Participants will wear these devices for 3 months.
  Interventions: Device: Fitbit Inspire 2; Device: Abbott Freestyle Libre 3
- Standard care (No Intervention): The control group will be given the standard recommendations that all patients completing cardiac rehabilitation receive.

INTERVENTIONS:
Device: Fitbit Inspire 2 — A smartwatch (Fitbit Inspire 2) with its respective app will be worn by the patients in the intervention group for 3 months.
  Arms: Wearing a smartwatch and glucose measuring device
Device: Abbott Freestyle Libre 3 — A continuous glucose measuring device (Abbott Freestyle Libre 3) with its respective app will be worn by the patients in the intervention group for 3 months.
  Arms: Wearing a smartwatch and glucose measuring device

SUMMARY:
The study aims to assess the effect of smart watches and continuous glucose measuring devices on cardiovascular risk factors.

DETAILED DESCRIPTION:
Within a period of 4 months 100 patients will be recruited and randomised to the intervention or control arm (1:1) for a duration of 3 months. Randomisation will be stratified by age, sex, BMI, diabetes, blood pressure, and duration after finishing cardiac rehabilitation. Patients randomised to the intervention arm will be given a smart watch as well as a continuous blood glucose measurement device with detailed instructions. At baseline and at the end of the study questionnaires will be answered and anthropomorphic measurements attained. Blood samples will be drawn at baseline and after an intervention period of 3 months in all subjects. Additional data on sleep, temperature, heart rate (resting and exercise), breathing rate, activity and exercise, oxygen saturation and daily weight will be collected through the Fitbit web application programming interface (API).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Completed outpatient cardiac rehabilitation
* Diagnosis of coronary heart disease
* Access to a smartphone for the duration of the study
* 18 years or older on the date of consent

Exclusion Criteria:

* Diseases which limit physical activity including angina with incomplete revascularisation, arrhythmogenic cardiomyopathy, stroke with residual disease, and major orthopaedic disorders
* Known or suspected non-compliance
* Inability to follow the procedures of the investigation, e.g., due to language problems, psychological disorders, dementia, etc. of the subject
* Diabetic patients receiving insulin therapy
* Lack of proficiency with smart phone/watch
* Current participation in any other clinical trial, which may confound the results of this trial.
* NYHA (New York Heart Association) class III or IV congestive heart failure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in cardiovascular risk factor score blood pressure | at baseline and after 3 month
  For the risk factor blood pressure 0 to 2 points will be awarded. 2 points will be rewarded if the patient reaches the goals according to ESC (European Society of Cardiology) -Guidelines where applicable, 1 point if the patient reaches the goal partially and 0 if the patient does not reach the goal.
  Goals according to ESC Guidelines:
  Systolic 120-130 mmHg (18-69y.) Systolic < 140 mmHg (70y.) Diastolic < 80 mmHg (all ages)
  Points according to goals:
  2 = age related SBP (systolic blood pressure) & DBP (diastolic blood pressure) goals
  1 = < 140 mmHg, > 130 mmHg 18-69yr. or < 140 mmHg and > 90 mmHg DBP >70yr 0 = SBP > 140 mmHg
Change in cardiovascular risk factor score LDL | at baseline and after 3 month
  For the risk factor LDL 0 to 2 points will be awarded. 2 points will be rewarded if the patient reaches the goals according to ESC-Guidelines where applicable, 1 point if the patient reaches the goal partially and 0 if the patient does not reach the goal.
  Goals according to ESC Guidelines:
  LDL <1.4 mmol/l and 50% reduction from baseline
  Points according to goals:
  2 = < 1.4 mmol/l
  1 = < 1.8 mmol/l 0 = > 1.8 mmol/l
Change in cardiovascular risk factor score HbA1c | at baseline and after 3 month
  For the risk factor HbA1c 0 to 2 points will be awarded. 2 points will be rewarded if the patient reaches the goals according to ESC-Guidelines where applicable, 1 point if the patient reaches the goal partially and 0 if the patient does not reach the goal.
  Goals according to ESC Guidelines:
  DM (diabetes mellitus) HbA1c < 7.0% or < 6.5% in recent diagnosis No DM < 5.7% (cut-off prediabetes)
  Points according to goals:
  2 = < 5.7 %
  1 = 5.7 - 6.5 % 0 = > 6.5 %
Change in cardiovascular risk factor score BMI | at baseline and after 3 month
  For the risk factor BMI 0 to 2 points will be awarded. 2 points will be rewarded if the patient reaches the goals according to ESC-Guidelines where applicable, 1 point if the patient reaches the goal partially and 0 if the patient does not reach the goal.
  Goals according to ESC Guidelines:
  BMI 20-25 kg/m2 AC (Abdominal circumference) < 102 (men) < 88 (women) WHR (waist to hip ratio) 0.75-0.9 men & 0.70-0.85 women
  Points according to goals:
  2 = BMI and AC in range
  1 = only BMI or AC in range 0 = nothing in range
Change in cardiovascular risk factor score physical activity | at baseline and after 3 month
  For the risk factor physical activity 0 to 2 points will be awarded. 2 points will be rewarded if the patient reaches the goals according to ESC-Guidelines where applicable, 1 point if the patient reaches the goal partially and 0 if the patient does not reach the goal.
  Goals according to ESC Guidelines:
  > 150min/week moderate PA (mPA), better 300min/week (self-reported) or > 75min/week vigorous PA (vPA), better 150min/week (self-reported)
  Points according to goals:
  2 = > 300 min. mPA or > 150 min. vPA
  1 = > 150 min. mPA or > 75 min. vPA 0 = < 150 min. mPA or < 75 min. vPA Or mix or mPA and vPA respectively
Change in cardiovascular risk factor score nutrition | at baseline and after 3 month
  For the risk factor nutrition 0 to 2 points will be awarded. 2 points will be rewarded if the patient reaches the goals according to ESC-Guidelines where applicable, 1 point if the patient reaches the goal partially and 0 if the patient does not reach the goal.
  Goals according to ESC Guidelines:
  ≥ 5 portions fruit/vegetables a day Unsalted nuts ≥ 3x/week Reduction in saturated fats
  Points according to goals:
  2 = 5/day OR 4/day + nuts 3x/week + reduction in saturated fats
  1 = 4/day OR 3/day + nuts 3x/week + reduction in saturated fats 0 = < 4/day
Change in cardiovascular risk factor score smoking | at baseline and after 3 month
  For the risk factor smoking 0 or 3 points will be awarded.
  Points according to goals:
  Smoking (yes/no) 3 = no 0 = yes

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gerrit van der Stouwe, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland